CLINICAL TRIAL: NCT04497701
Title: A Multi-center, Open-label, Randomized Controlled Study to Evaluate the Efficacy and Safety of the Prophylactic Use of Pegylated Recombinant Human Granulocyte Colony Stimulating Factor After Chemotherapy in Children With Hematological Malignancies
Brief Title: Evaluate the Efficacy and Safety of the Prophylactic Use of PEG-rhG-CSF in Children With Hematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Collaborators: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-JYL-CHIL-01
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Lymphoma; Leukemia
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEG-rhG-CSF group (Experimental): Patients received subcutaneous injection of PEG-rhG-CSF(Jinyouli®)24~72 hours after the end of chemotherapy, 100µg/kg, once in each chemotherapy cycle.
  Interventions: Drug: PEG-rhG-CSF group
- rhG-CSF group (Active Comparator): Patients received subcutaneous injection of rhG-CSF 24~72 hours after the end of chemotherapy, 100µg/kg/d, and stop using it until the ANC value exceeds the lowest value for 2 consecutive days> 0.5×10^9/L.
  Interventions: Drug: rhG-CSF group

INTERVENTIONS:
Drug: PEG-rhG-CSF group — Patients received a single dose of 100 ug/kg of PEG-rhG-CSF（Jinyouli®）, on the basis of actual body weight. Peg-rhG-CSF can be used prophylactically only when the interval between two chemotherapy regimens is no less than 12 days.
  Arms: PEG-rhG-CSF group
Drug: rhG-CSF group — Patients received 5μg/kg/d of rhG-CSF, on the basis of actual body weight.
  Arms: rhG-CSF group

SUMMARY:
The incidence of infectious complications in hematological malignancies is higher than that in children with solid tumors, which may be related to the type and dose intensity of chemotherapy regimens used in hematological tumors. The treatment of childhood cancer has changed in the past few decades: intensive treatment and good supportive treatment can improve the 5-year survival rate of children. The aim of this study was to evaluate the efficacy and safety of prophylactic use of pegylated recombinant human granulocyte colony-stimulating factor (PEG-rhG-CSF) after chemotherapy in children with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Under the age of 18, no gender limit;
2. Children with hematological malignancies, leukemia or lymphoma, diagnosed by bone marrow pathology or cytology;
3. The prophylactic use of PEG-rhG-CSF or rhG-CSF after chemotherapy is intended to prevent neutropenia, and the chemotherapy regimen must meet the interval between two chemotherapy sessions at least 12 days;
4. The effect of chemotherapy in leukemia patients was complete remission, while that in lymphoma patients was complete remission or partial remission;
5. The expected survival time is more than 8 months;
6. Liver and kidney function: Liver function: total bilirubin (TBIL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal value, or≤5 times the upper limit of normal value when there is liver metastasis; renal function test: serum creatinine (Cr) ≤ 1.5 times the upper limit of normal value;
7. Eastern Cooperative Oncology Group(ECOG) performance status(PS) <2;
8. The subjects had good mental consciousness, and the subject's legal guardian must sign an informed consent form;
9. Researchers believe that the subject can benefit;

Exclusion Criteria:

1. Severe internal organ dysfunction;
2. Those who used other test drugs of the same kind or accepted other clinical trials within 4 weeks before enrollment;
3. Allergy to PEG-rhG-CSF, rhG-CSF and other preparations or proteins expressed by Escherichia coli;
4. Researchers determine unsuited to participate in this trial.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 139 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia (FN) | From date of randomization until the date of the study completion, up to 24 weeks.
  ANC<0.5×10^9/L or ANC (0.5-0.9)×10^9/L, and predicted to drop to ≤0.5×10^9/L in the next 48 hours, and the oral cavity temperature is ≥38.3℃ or ≥38.0℃ for more than 1 hour.

SECONDARY OUTCOMES:
Duration of febrile neutropenia | From date of randomization until the date of the study completion, up to 24 weeks.
  Defined as days when the FN occurs to the time when FN disappears.
Incidence and duration of grade IV neutropenia (ANC<0.5×10^9/L) | From date of randomization until the date of the study completion, up to 24 weeks.
  Grade IV neutropenia is defined as the absolute neutrophil count(ANC)<0.5×10^9/L; Duration of grade IV neutropenia is defined as days when the ANC<0.5×10^9/L occurs to the time when the ANC≥0.5×10^9/L
Recovery time of grade IV neutropenia | From date of randomization until the date of the study completion, up to 24 weeks.
  Time from the first day of chemotherapy to ANC≥0.5×10^9/L
Dynamic curve of absolute neutrophil count (ANC) | From date of randomization until the date of the study completion, up to 24 weeks.
  Dynamic changes of ANC after chemotherapy
Hospital stay | From date of randomization until the date of the study completion, up to 24 weeks.
  Number of days the patient was hospitalized
Incidence of infection | From date of randomization until the date of the study completion, up to 24 weeks.
  Incidence of various infections
Dose adjustment of chemotherapy or delay of chemotherapy | From date of randomization until the date of the study completion, up to 24 weeks.
  Dose adjustment of chemotherapy is defined as incidence of the reduction of planned dose of chemotherapy；Chemotherapy delay is defined as the delay in starting the next planned chemotherapy for more than 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Zhai, Doctor, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China